CLINICAL TRIAL: NCT01700231
Title: Monitoring Plasma and Hemodynamic Markers in Patients Undergoing Liver Resection to Identify Pathophysiological Mechanisms and Predict Clinical Outcome
Brief Title: Plasma and Hemodynamic Markers During Hepatectomy
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Edith Fleischmann, Clinical Professor, Medical University of Vienna
Other Study IDs: HVPG/Liver Regeneration Study
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hepatorenal Syndrome, Liver Regeneration
Keywords: hepatorenal syndrome, liver regeneration, liver dysfunction
MeSH Terms: conditions — Hepatorenal Syndrome; Liver Diseases | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — perioperative plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver resection ,Liver Dysfunction: 100 patients will be monitored perioperatively, in a subset of 40 patients hepatic venous pressure gradient will be monitored
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Liver resection — Liver resection of patient with neoplastic hepatic tumors

SUMMARY:
Introduction Liver resection is considered the only curative treatment option for mCRC patients without extrahepatic disease and is accepted practice. Despite substantial improvements in surgical techniques, postoperative morbidity and mortality remain an important concern after major resections. Complications of liver resection, although rare, include liver failure and acute kidney injury as indicated by oliguria and increased serum creatinine. The underlying pathophysiological pathways of post-operative renal alteration following liver resection is an increase in portal venous pressure, based on observations in animal models or small cohorts. The corpus of data is derived from patients with liver cirrhosis and subsequent hepatorenal syndrome. These data are limited since cirrhosis cannot distinguish between metabolic changes, portal hypertension and impaired liver function in the elucidation of the pathogenesis of renal alterations. Liver resection is therefore a potent model to evaluate the impact of portal hypertension on the kidney despite stable liver function.

The most significant factor determining morbidity and mortality following hepatectomy is the ability of the remnant liver to regenerate. In this context, several growth factors were shown to regulate the highly orchestrated process of liver regeneration (LR).

Hypothesis The investigators will therefore test the hypothesis that liver resection leads to a sustained increase of portalvenous pressure with a subsequent episode of oliguric renal impairment, correlating with the quantity of resected liver.

Furthermore, the investigators will examine the relationship between postoperative liver regeneration and circulating growth factor levels in patients undergoing hepatectomy. Based on the preclinical data the investigators hypothesize that a circulating growth factor levels will be associated with delayed liver regeneration, an increased incidence of postoperative liver dysfunction and concomitant worse clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neoplastic liver tumors undergoing elective hepatectomy.

Exclusion Criteria:

* Non elective hepatic surgery, preoperative HVPG > 10 mmHG, preoperative renal failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with neoplastic liver tumors undergoing hepatectomy.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-10; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Perioperative blood parameters and HVPG | 90 postoperative days
  Time course and predictive potential of blood parameter and HVPG in patients undergoing liver resection. Clinical outcome parameters are postoperative morbidity, mortality and liver dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Edith Fleischmann, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- General Hospital Vienna, Vienna, Austria

REFERENCES:
- [Derived] Starlinger P, Pereyra D, Haegele S, Braeuer P, Oehlberger L, Primavesi F, Kohler A, Offensperger F, Reiberger T, Ferlitsch A, Messner B, Beldi G, Staettner S, Brostjan C, Gruenberger T. Perioperative von Willebrand factor dynamics are associated with liver regeneration and predict outcome after liver resection. Hepatology. 2018 Apr;67(4):1516-1530. doi: 10.1002/hep.29651. Epub 2018 Feb 27. PMID 29140542
- [Derived] Padickakudy R, Pereyra D, Offensperger F, Jonas P, Oehlberger L, Schwarz C, Haegele S, Assinger A, Brostjan C, Gruenberger T, Starlinger P. Bivalent role of intra-platelet serotonin in liver regeneration and tumor recurrence in humans. J Hepatol. 2017 Dec;67(6):1243-1252. doi: 10.1016/j.jhep.2017.08.009. Epub 2017 Aug 24. PMID 28842294
- [Derived] Pereyra D, Offensperger F, Klinglmueller F, Haegele S, Oehlberger L, Gruenberger T, Brostjan C, Starlinger P. Early prediction of postoperative liver dysfunction and clinical outcome using antithrombin III-activity. PLoS One. 2017 Apr 13;12(4):e0175359. doi: 10.1371/journal.pone.0175359. eCollection 2017. PMID 28406940
- [Derived] Starlinger P, Assinger A, Haegele S, Wanek D, Zikeli S, Schauer D, Birner P, Fleischmann E, Gruenberger B, Brostjan C, Gruenberger T. Evidence for serotonin as a relevant inducer of liver regeneration after liver resection in humans. Hepatology. 2014 Jul;60(1):257-66. doi: 10.1002/hep.26950. PMID 24277679